CLINICAL TRIAL: NCT05173350
Title: One-Year Impact Evaluation of Retaining Employment and Talent After Injury/Illness Network (RETAIN) Kentucky
Brief Title: RETAIN Kentucky Impact Evaluation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mathematica Policy Research, Inc. (Other)
Collaborators: Social Security Administration, The United States (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RTN-KY; OD-36364-21-75-4-21 (Other Grant/Funding Number: SSA)
Record Dates: First submitted 2021-11-05; First posted 2021-12-29 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2021-11

CONDITIONS: Disability
Keywords: disability; employment; unemployment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RETAIN Programming (Experimental): The experimental group receives the full set of RETAIN intervention activities.
  Interventions: Other: RETAIN KY
- Active Comparator (Active Comparator): The active comparator group does not receive the full set of RETAIN intervention activities.
  Interventions: Other: Active Comparator

INTERVENTIONS:
Other: RETAIN KY — The experimental group receives a combination of medical provider services, stay-at-work (SAW)/return-to-work (RTW) coordination services, and other SAW/RTW services. Services offered by the project include individualized intensive vocational services from RETAIN RTW Coordinators, with an emphasis on assistive technology, universal design, and peer support. The project provides training on SAW/RTW best practices and RETAIN, as well as financial incentives to health care professionals. The treatment group is eligible to receive the full set of RETAIN intervention activities.
  Arms: RETAIN Programming
Other: Active Comparator — Those in the active comparator arm continue to receive medical services. A RTW coordinator creates a RTW plan with the enrollee and refers them to existing resources. The RTW coordinator works with enrollees for 2.5 hours total.
  Arms: Active Comparator

SUMMARY:
The Retaining Employment and Talent after Injury/Illness Network (RETAIN) demonstration is a collaborative effort between the U.S. Department of Labor (DOL) and the Social Security Administration (SSA) to improve employment outcomes for individuals who experience injuries or illnesses that put them at risk of exiting the labor force and relying on disability programs and other public supports in the long term. RETAIN projects include a combination of medical provider services, stay-at-work/return-to-work (SAW/RTW) coordination services, and other SAW/RTW services. This evaluation will focus on The Kentucky Education and Workforce Development Cabinet's implementation of "RETAIN KY" statewide. The evaluation will document how the project is implemented, describe enrollees, estimate the project's impacts on enrollees' outcomes, and assess whether the benefits outweigh the costs.

DETAILED DESCRIPTION:
SSA contracted with Mathematica to conduct an independent evaluation of RETAIN Kentucky. Under the RETAIN model medical providers receive training and incentives to use occupational health best practices. The state agency also coordinates SAW/RTW services for the enrollee, fosters communication among RETAIN stakeholders about the treatment enrollee returning to work, and monitors the enrollee's medical and employment progress. RETAIN Kentucky also provides individualized intensive vocational services from RETAIN RTW Coordinators, with an emphasis on assistive technology, universal design, and peer support.

Kentucky uses a multi-method approach toward recruitment that includes referrals from medical providers, employers, Office of Vocational Rehabilitation, workforce and disability management organizations, community partners, and word of mouth. A return-to-work (RTW) coordinator conducts intake, determines enrollees' eligibility, and randomly assigns each enrollee to either a treatment group that is eligible to receive the full set of RETAIN intervention activities or a control group that is not. The evaluation team then compares the outcomes of the two groups and gathers evidence on how each RETAIN project shaped the outcomes of enrollees who were eligible for its services, regardless of whether they participated in those services. Data sources include enrollment data, surveys, administrative records, program data, and qualitative data.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are at risk of exiting the workforce due to non-work-related illness of injury
* Individuals who are employed or have been employed within the last 12 months and made at least $1,000 in one of those months
* Individuals who reside in the Kentucky
* Individuals must not have applied for or be receiving federal disability benefits including SSDI and SSI within the last 5 years

Exclusion Criteria:

* Individuals who are do not have a non-work-related illness or injury that puts them at risk of exiting the workforce
* Individuals who unemployed or have not been employed within the last 12 months
* Individuals who have not made at least $1,000 in the past 12 months
* Individuals who do not reside in the Kentucky
* Individuals who have applied for or be receiving federal disability benefits including SSDI and SSI within the last 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3200 (Estimated)
Dates: Start 2021-10-18 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Share of enrollees employed in the fourth quarter after enrollment | Measured over the three months in the fourth quarter after enrollment
  Share of enrollees employed in the fourth quarter after enrollment obtained from state unemployment insurance wage records. These files include individual-level wage records for six quarters surrounding enrollment in the study, including the quarter prior to enrollment, the quarter of enrollment, and four post-enrollment quarters.
Enrollee earnings in the fourth quarter after enrollment | Measured over the three months in the fourth quarter after enrollment
  Sum of enrollee earnings in the fourth quarter after enrollment obtained from state unemployment insurance wage records. These files include individual-level wage records for six quarters surrounding enrollment in the study, including the quarter prior to enrollment, the quarter of enrollment, and four post-enrollment quarters.
Share of enrollees that applied for SSDI or SSI during the 12 months after enrollment | Measured in the 12 months after enrollment
  Share of enrollees that applied for SSDI or SSI during any of the 12 months after enrollment obtained from SSA program data. These files include detailed information about Social Security Disability Insurance (SSDI) and Supplemental Security Income (SSI) applications SSDI and SSI awards, SSDI and SSI benefit amounts and enrollee characteristics (for enrollees who have ever applied for SSA program benefits)

CONTACTS AND LOCATIONS:
Overall Officials: Jill Berk, PhD, Principal Investigator — Mathematica Policy Research, Inc.
Locations (1):
- Human Development Institute, University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No